CLINICAL TRIAL: NCT06918457
Title: A Clinical Trial With a Self-controlled, Multicenter, Pediatric EEG Intelligent Analysis System to Assist in Diagnosis
Status: Not yet recruiting | Type: Observational
Sponsor: Kunming Children's Hospital (Other)
Responsible Party: Principal Investigator, Xiaomei Liu, Professor, Kunming Children's Hospital
Other Study IDs: 2024-03-278-K01
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: AI EEG analysis system — The first stage, physicians independently diagnose pediatric epilepsy with EEG; the second stage, Artificial intelligence EEG analysis system assisted physicians to diagnose pediatric epilepsy

SUMMARY:
A diagnostic accuracy study on Artificial intelligence EEG analysis system assisted doctors to diagnose pediatric epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years old
* Children with suspected epilepsy

Exclusion Criteria:

* During EEG monitoring, the patients had other serious neurological diseases and mental diseases concurrently
* Used medication that affect EEG data within 3 weeks, such as sedatives and anti-epileptic medications
* Substandard data quality, such as data lack of key records, electrode connection discontinuity, insufficient recording time, or the presence of serious artifacts
* Incomplete or missing data
* Equipment or operational abnormalities, data for which EEG monitoring has not been performed continuously

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children aged < 18 years old with suspected epilepsy who need EEG examination
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-03 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the coincidence rate between doctors' independent diagnosis and the diagnosis recommended by the AI system. | Within 48 hours after the completion of EEG monitoring
  The reference standard is the EGG interpreted by 3 clinicians who had attended the uniformly training program and had more than 5 years of experience in diagnosing epilepsy in children.

SECONDARY OUTCOMES:
To evaluate the diagnostic efficiency of clinicians at two-stage | Immediately after the end of EEG interpretation
  The time taken by physicians to interpret EEG independently and with the aid of AI was measured.

IPD SHARING:
Plan to Share IPD: No